CLINICAL TRIAL: NCT05581914
Title: The Effectiveness of the MY LIFE Treatment for Adolescents With Behavioral Problems: a Group Randomized Controlled Trial and Qualitative Analyses of Client Evaluations.
Brief Title: Effectiveness of the MY LIFE Treatment for Adolescents With Behavioral Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Helena Oldenhof, Doctor Helena Oldenhof (PhD) Sponsor-Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT MY LIFE
Record Dates: First submitted 2022-10-05; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Behavior Problem
Keywords: Behavioral problems; Transdiagnostic treatment; Adolescents; Self-worth; Hope; Seeking support; Peer expert
MeSH Terms: conditions — Mental Disorders; Problem Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Care as Usual and the MY LIFE treatment
  Interventions: Other: MY LIFE treatment
- Waitinglist Control group (Active Comparator): Care as Usual
  Interventions: Other: Care as Usual

INTERVENTIONS:
Other: MY LIFE treatment — The MY LIFE is a group treatment consisting of 5 workshops, for adolescents with a low motivation for mental health treatment. It aims to increase self- worth, hope for the future and seeking social support through exercises by using music and lyrics and other creative exercises to engage adolescents. The MY LIFE treatment also uses methods that stem from psychodynamic, cognitive behavioral, and solution focused theories. The therapeutic attitude is based on client-centered therapy of Rogers, which includes a genuine, positive regard and empathic understanding, focusing on the inner strength and growth potential of a person. Adolescents are never forced to participate during the workshops, merely encouraged.
  The core of the treatment is: the adolescent decides
  Arms: Treatment group
Other: Care as Usual — The care as usual the adolescents receives
  Arms: Waitinglist Control group

SUMMARY:
Objective This study examines the effects of the MY LIFE treatment, a group intervention aiming to increase hope, self-worth and social support seeking in adolescents with behavioral problems in mental health care.

Method This study is a group randomized controlled trial to determine whether MY LIFE is effective, by comparing care as usual with care as usual plus the MY LIFE treatment. Groups of adolescents (N= 50 per arm, Age= 14-20) with behavioral problems will be randomly assigned to either the care as usual condition or the care as usual plus the MY LIFE treatment condition. The second part of the study is focused on the subjective evaluation of the intervention by the adolescents, using qualitative research methods.

Results Primary outcomes of the RCT are hope, self-worth, and seeking social support. As secondary outcomes emotional and behavioral symptoms are assessed. The second part of the study analyses the subjective evaluation of the MY LIFE treatment.

DETAILED DESCRIPTION:
Treating adolescents with behavioral problems without motivation for change in youth mental healthcare is a challenge, and group interventions targeting these adolescents show low effectiveness. This seems even more pronounced in girls. Most interventions focus on behavioral change and include parental involvement. The MY LIFE treatment was designed to provide a treatment based on the needs of adolescents. A good working alliance is essential in treatment. For instance, the alliance between girls and staff in residential care, predicts treatment success, and a weak working alliance is associated with more behavioral problems. According to evaluations of successful treatments at our mental health department for complex behavioral problems, adolescents value the concepts of hope, self-worth and seeking support as well. Therefore, these concepts, as well as the working alliance, were key elements in the development of the MY LIFE treatment.

Hope This study uses Snyder's definition: "hope is a positive motivational state that is based on an interactively derived sense of successful (a) agency (goal-directed energy) and (b) pathways (planning to meet goals)" . The relevance of the concept of hope for adolescents with mental health problems has been widely studied. For instance, hope makes children resilient to adverse life events. The prevalence of adverse life events is high in children and adolescents with behavioral problems, which emphasizes the importance of addressing this concept in interventions for these adolescents.

Self-worth In this study self-worth is defined as a person's subjective evaluation of his or hers own worth. Low self-worth is related to aggression and antisocial behavior, and addressing this concept in the treatment of behavioral problems of adolescents may help to reduce aggressive and antisocial behavior.

Seeking support The definition of seeking support used here, is "having an active coping style when facing problems or stressful situations" . An active coping style leads to a greater well-being in adolescents. Therefore, teaching them an active coping style, such as seeking support, is important in an attempt to reduce behavioral problems and to foster well-being in adolescents witt behavioral problems. These findings suggest coping should be a target for intervention.

These three concepts are interrelated; active coping such as seeking support is related to more self-worth and vice versa: better social relationships lead to more self-worth. Furthermore, studies show that self- worth mediates the association of hope with life satisfaction.

Objectives and research questions

The study aims to examine the effectiveness of the MY LIFE treatment, answering the following questions:

1. Do adolescents with behavioral problems (age 14-20) receiving MY LIFE in addition to care as usual, have more hope after the treatment, compared to the adolescents in the waitinglist control group receiving only care as usual?
2. Do adolescents with behavioral problems (age 14-20) receiving MY LIFE in addition to care as usual have a higher level of self-worth after the treatment, compared to the waitinglist control group receiving only care as usual?
3. Do adolescents with behavioral problems (age 14-20) receiving MY LIFE in addition to care as usual seek more support after the treatment compared to the waitinglist control group receiving only care as usual?
4. Do adolescents with behavioral problems (age 14-20) have more hope, a higher level of self-worth and seek more support after receiving MY LIFE, in comparison to pre-treatment?

   Secondary, this study focuses on the question:
5. Is there a change in behavioral and emotional symptoms (emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, prosocial behavior, disruptive behavior, anger) in adolescents with behavioral problems (age 14-20) receiving MY LIFE in addition to care as usual, as compared to adolescents in the waitinglist control group receiving only care as usual? The second part of this study uses a structured interview to assess the subjective evaluation of the treatment by the adolescents.

Method Trial management The trial is funded by KFZ-J (Kwaliteit Forensische Zorg Jeugd) and led by a team of researchers and clinicians from the AmsterdamUMC and Levvel (youth mental health care).

Study design The study is a group randomized controlled trial, comparing Care As Usual (CAU) plus the MY LIFE treatment with a waitinglist control group receiving only CAU. The study procedure is depicted in figure 1. All adolescents and a chosen caretaker (CC) by the adolescent, will fill in questionnaires during a baseline assessment (T0). Six weeks later all adolescents and the CC will again fill in questionnaires during a post-measurement (T1). The waitinglist control group will receive the MY LIFE treatment after T1 and an additional post-measurement will be done after they have received the treatment (T2). All adolescents will be asked to fill in the questionnaires again 1 year after T0 (T3).

The Medical Ethics Review Committee of VU University Medical Center (METC) has reviewed the study protocol and concluded that the Medical Research Involving Human Subjects Act (WMO) does not apply to this study. The Medical Ethics Review Committee of VU University Medical Center is registered with the US Office for Human Research Protections (OHRP) as IRB00002991. The FWA number assigned to VU University Medical Center is FWA00017598.

Data management Since this is the first study on the MY LIFE treatment, and this treatment is different than interventions used in this population, it is difficult to estimate the expected effect and also the required sample size. Furthermore, previous studies in similar populations have demonstrated a large variety in effectsized of CBT-based interventions, ranging from small (d=0.33) to large (d=0.98) effects. To calculate the sample size for this study we used G* Power, with an estimation effect of (d=0.5), a power of β=0.8 and an ICC=0.6 to correct for dependency between the repeated measures. This resulted in an N of 50 adolescents per arm (in total N= 100) for this RCT.

A group randomized controlled trial will be performed to evaluate the effect of the intervention. All groups will receive care as usual within their youth care facility. The treatment group will also receive the MY LIFE treatment. Castor, a data management software program, will be used to store the data. To analyse the data a multilevel model with a three level structure (repeated measures are clustered within participants, and participants are clustered within groups) will be used via SPSS (Statistical Package for the Social Sciences). Analyses will be performed twice: once based on intention-to-treat (we consider this our primary analysis), and once including only those adolescents who completed the intervention. Missing data is taken into account by the multilevel analyses. Outliers deviating 3SD from the mean will be excluded.

The qualitative data will be analysed using ATLAS.ti.

ELIGIBILITY:
Inclusion Criteria:

Adolescent is referred for behavioral problems

Exclusion Criteria:

School level is below BL (a school level in the Dutch school system)

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
JIJ questionnaire | For the Treatment arm: at the first intake, 7 weeks after the intake, one year after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment, one year after intake
  Hope/ Self-worth/ Seeking support Self report
CHS (Children Hope Scale) | For the Treatment arm: at the first intake, 7 weeks after the intake, one year after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment, one year after intake
  Hope Self report
BSCI-Y (Beck Self- Concept Inventory for Youth) | For the Treatment arm: at the first intake, 7 weeks after the intake, one year after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment, one year after intake
  Self-worth Self report
UCL (S) Utrechtse Coping List Social support | For the Treatment arm: at the first intake, 7 weeks after the intake, one year after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment, one year after intake
  Seeking support Self Report
JIJ questionnaire BA | For the Treatment arm: at the first intake, 7 weeks after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment.
  Hope/ Self -worth/ Seeking support. Form is filled in by a caregiver chosen by the adolescent.
KLAD (Klachtenlijst Adolescenten) subscale self-worth | For the Treatment arm: at the first intake, 7 weeks after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment.
  Self- Worth Form is filled in by caregiver chosen by the adolescent.
KLAD (Klachtenlijst Adolescenten) subscale social support | For the Treatment arm: at the first intake, 7 weeks after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment.
  Seeking support Form is filled in by caregiver chosen by the adolescent

SECONDARY OUTCOMES:
SDQ (Strengths and Difficulties Questionnaire) | For the Treatment arm: at the first intake, 7 weeks after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment.
  Emotional symptoms Conduct problems Hyperactivity/inattention Peer relationship problems Prosocial behavior Self report
BDBI-Y (Beck Disruptive Behavior Inventory for Youth) | For the Treatment arm: at the first intake, 7 weeks after the intake, one year after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment, one year after intake
  Disruptive behavior self report
BANI-Y (Beck Anger Inventory for Youth) | For the Treatment arm: at the first intake, 7 weeks after the intake, one year after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment, one year after intake
  Anger self report
Workshop evaluation designed for the purpose of this study | per workshop so every week during the treatment, 5 times
  Client satisfaction regarding workshop with three smilies. Self report
Strengths and Difficulties Questionnaire (SDQ) for parents or teachers | For the Treatment arm: at the first intake, 7 weeks after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment.
  Emotional symptoms, Conduct problems, Hyperactivity/Inattention, Peer relationship problems, Prosocial behavior
KLAD (Klachtenlijst Adolescenten) subscale emotional difficulties | For the Treatment arm: at the first intake, 7 weeks after the intake. For the waiting list control group: at the intake, 7 weeks after intake, 7 weeks later after treatment.
  Emotional difficulties. Form is filled in by a caregiver chosen by the adolescent

OTHER OUTCOMES:
Evaluation of the MY LIFE treatment | 6 weeks after start treatment
  evaluation by the adolescents of the MY LIFE treatment

CONTACTS AND LOCATIONS:
Overall Officials: T.J. Dekkers, PhD, Study Chair — AmsterdamUMC; J.W.R. Twisk, Prof.Dr, Study Chair — AmsterdamUMC; A. Popma, Prof.Dr, Study Director — AmsterdamUMC
Locations (1):
- Levvel, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
No sharing of data after the study. Merely for use in this particular study.

REFERENCES:
- [Background] Ayotte, M. H., Lanctôt, N., & Tourigny, M. (2016). How the working alliance with adolescent girls in residential care predicts the trajectories of their behavior problems. Residential Treatment for Children & Youth, 33(2), 135-154. https://doi.org/10.1080/0886571x.2016.1175994
- [Background] Barendregt CS, Van der Laan AM, Bongers IL, Van Nieuwenhuizen C. Adolescents in secure residential care: the role of active and passive coping on general well-being and self-esteem. Eur Child Adolesc Psychiatry. 2015 Jul;24(7):845-54. doi: 10.1007/s00787-014-0629-5. Epub 2014 Oct 18. PMID 25325990
- [Background] Barendregt CS, van der Laan AM, Bongers IL, van Nieuwenhuizen C. Longitudinal Relation Between General Well-Being and Self-Esteem. Int J Offender Ther Comp Criminol. 2016 Dec;60(16):1836-1855. doi: 10.1177/0306624X15588773. Epub 2016 Jul 28. PMID 26063543
- [Background] Baxter MA, Hemming EJ, McIntosh HC, Hellman CM. Exploring the Relationship Between Adverse Childhood Experiences and Hope. J Child Sex Abus. 2017 Nov-Dec;26(8):948-956. doi: 10.1080/10538712.2017.1365319. Epub 2017 Aug 31. PMID 28857691
- [Background] Boeije, H. (2016). Analyseren in kwalitatief onderzoek: Denken en doen. Boom Lemma.
- [Background] Dam, C. V., Nijhof, K. S., Scholte, R. H. J., & Veerman, J. W. (2010). Evaluatie nieuw zorgaanbod: Gesloten jeugdzorg voor jongeren met ernstige gedragsproblemen: Eindrapport
- [Background] Donnellan MB, Trzesniewski KH, Robins RW, Moffitt TE, Caspi A. Low self-esteem is related to aggression, antisocial behavior, and delinquency. Psychol Sci. 2005 Apr;16(4):328-35. doi: 10.1111/j.0956-7976.2005.01535.x. PMID 15828981
- [Background] Du, H., Bernardo, A. B., & Yeung, S. S. (2015). Locus-of-hope and life satisfaction: The mediating roles of personal self-esteem and relational self-esteem. Personality and Individual Differences, 83, 228-233. https://doi.org/10.1016/j.paid.2015.04.026
- [Background] Frydenberg E, Lewis R. Relations among well-being, avoidant coping, and active coping in a large sample of Australian adolescents. Psychol Rep. 2009 Jun;104(3):745-58. doi: 10.2466/PR0.104.3.745-758. PMID 19708401
- [Background] Granski M, Javdani S, Anderson VR, Caires R. A Meta-Analysis of Program Characteristics for Youth with Disruptive Behavior Problems: The Moderating Role of Program Format and Youth Gender. Am J Community Psychol. 2020 Mar;65(1-2):201-222. doi: 10.1002/ajcp.12377. Epub 2019 Aug 26. PMID 31449683
- [Background] Harris MA, Orth U. The link between self-esteem and social relationships: A meta-analysis of longitudinal studies. J Pers Soc Psychol. 2020 Dec;119(6):1459-1477. doi: 10.1037/pspp0000265. Epub 2019 Sep 26. PMID 31556680
- [Background] Horvath AO, Luborsky L. The role of the therapeutic alliance in psychotherapy. J Consult Clin Psychol. 1993 Aug;61(4):561-73. doi: 10.1037//0022-006x.61.4.561. PMID 8370852
- [Background] McLeod BD. Relation of the alliance with outcomes in youth psychotherapy: a meta-analysis. Clin Psychol Rev. 2011 Jun;31(4):603-16. doi: 10.1016/j.cpr.2011.02.001. Epub 2011 Mar 17. PMID 21482319
- [Background] Muarifah A, Mashar R, Hashim IHM, Rofiah NH, Oktaviani F. Aggression in Adolescents: The Role of Mother-Child Attachment and Self-Esteem. Behav Sci (Basel). 2022 May 17;12(5):147. doi: 10.3390/bs12050147. PMID 35621444
- [Background] Peeters, J. (1994). Klachtenlijst voor adolescenten: KLAD (Complaintlist for Adolescents). Gedragstherapie, 27(2), 109-125.
- [Background] Riise EN, Wergeland GJH, Njardvik U, Ost LG. Cognitive behavior therapy for externalizing disorders in children and adolescents in routine clinical care: A systematic review and meta-analysis. Clin Psychol Rev. 2021 Feb;83:101954. doi: 10.1016/j.cpr.2020.101954. Epub 2020 Dec 7. PMID 33418192
- [Background] ROGERS CR. Significant aspects of client-centered therapy. Am Psychol. 1946 Oct;1(10):415-22. doi: 10.1037/h0060866. No abstract available. PMID 20280375
- [Background] Sanetti, L. M. H., Cook, B. G., & Cook, L. (2021). Treatment fidelity: What it is and why it matters. Learning Disabilities Research& Practice, 36(1), 5-11.
- [Background] Schreurs, P. J. P., Van de Willige, G., Tellegen, B., Brosschot, J. F., & Graus, G. M. H. (1993). De Utrechtse coping lijst: UCL: omgaan met problemen en gebeurtenissen. Harcourt Test Publ.
- [Background] Sheffler JL, Piazza JR, Quinn JM, Sachs-Ericsson NJ, Stanley IH. Adverse childhood experiences and coping strategies: identifying pathways to resiliency in adulthood. Anxiety Stress Coping. 2019 Sep;32(5):594-609. doi: 10.1080/10615806.2019.1638699. Epub 2019 Jul 9. PMID 31288568
- [Background] Twisk J, de Boer M, de Vente W, Heymans M. Multiple imputation of missing values was not necessary before performing a longitudinal mixed-model analysis. J Clin Epidemiol. 2013 Sep;66(9):1022-8. doi: 10.1016/j.jclinepi.2013.03.017. Epub 2013 Jun 21. PMID 23790725
- [Background] Twisk, J. W. R. (2021). Analysis of data from randomized controlled trials: A practical guide (1st ed. 2021). Springer.